CLINICAL TRIAL: NCT05869864
Title: Schools Championing Safe South Africa: An Intervention Engaging Teachers and Students in Adolescent Prevention of HIV Risk and Intimate Partner Violence
Brief Title: Schools Championing Safe South Africa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Caroline Kuo, Associate Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Schools Championing
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Prevention or Reduction of HIV Risk Behavior; Prevention or Reduction of Intimate Partner Violence

STUDY DESIGN:
Intervention Model Description: The primary goal of this study is to assess acceptability of the behavioral intervention in a small group of participants and to determine feasibility of the study design for a future fully-powered clinical trial. The secondary goal of this study is to evaluate under-powered directions of behavior change relating to prevention or reduction of HIV risk behavior and intimate partner violence.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Half of the participants in the pilot will receive the experimental behavioral intervention.
  Interventions: Behavioral: Schools Championing Safe South Africa
- Control (No Intervention): Half of the participants in the pilot will receive nothing, and serve as the control.

INTERVENTIONS:
Behavioral: Schools Championing Safe South Africa — The intervention consists of 2 parts - a poster campaign with social norms messages on violence and HIV risk, and 2 lessons in life orientation (a health curriculum delivered during school).
  Arms: Intervention

SUMMARY:
This study explores the acceptability and feasibility of a school-based intervention called Schools Championing Safe South Africa that engages teachers and students in an integrated approach for preventing risk behavior related to acquisition of HIV and perpetration of IPV among adolescents in South Africa. Teachers and students are agents of change who can transform the school social environment to promote HIV and IPV prevention behaviors for adolescents.

DETAILED DESCRIPTION:
Adolescence presents an ideal developmental transition period for an integrated intervention targeting prevention of HIV risk behaviors and intimate partner violence (IPV) including sexual violence. Adolescent boys in particular, are at high risk for HIV and perpetration of IPV. Yet, few behavioral interventions integrate HIV-IPV prevention and are tailored for the unique developmental needs of adolescent boys. Educational environments play a vital role in shaping behavioral choices among adolescent boys. Specifically, teachers and student peers serve as agents of change for adolescent boys' HIV and IPV prevention needs in four important ways. First, teachers and student peers influence community norms for appropriate adolescent male behaviors relating to dating, relationships, and sexual violence within the school ecology. Second, teachers and student peers have persistent contact with adolescents and thus, can play an influential role in adolescents' lives as role models for healthy norms. Third, teachers and student peers substantively motivate and reinforce protective behaviors relating to prevention of HIV and IPV. Fourth, teachers are ideally prepared to deliver age- and developmentally-tailored preventive interventions to adolescents because they are professionally trained to engage with adolescents in age and developmentally appropriate teaching. Despite the important role of teachers and student peers in promoting the health of adolescents, there are currently no HIV-IPV interventions in global priority settings for these epidemics that target teachers and student peers in school environments. In this study, we will develop and then investigate the acceptability and feasibility of Schools Championing Safe South Africa, an integrated HIV-IPV intervention where teachers and student peers engage adolescent boys in a developmentally-tailored approach to prevent adolescent HIV risk behavior and IPV using a social norms approach. Investigators work in South Africa, a country with the largest HIV epidemic and some of the highest rates of IPV in the world. This study explores the acceptability and feasibility of a school-based intervention called Schools Championing Safe South Africa that engages teachers and students in an integrated approach for preventing risk behavior related to acquisition of HIV and perpetration of IPV among adolescents in South Africa. Teachers and students are agents of change who can transform the school social environment to promote HIV and IPV prevention behaviors for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* identifies as boy
* 15-17 years of age inclusive
* attends school where study is occurring

Exclusion Criteria:

* unable to secure parental consent
* unable to secure parental consent child assent

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2025-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- South African Medical Research Council, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While teachers were exposed to the intervention (including the poster campaign), they were not the main target of the intervention.Thus, data on the primary outcomes of the study was not gathered from teachers.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 142 | 140
Completed | 142 | 140
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 142 | 140 | 282
Age, Categorical [Count of Participants; unit: Participants]
  Participants under 18 years: <=18 years | 142 | 140 | 282
  Participants under 18 years: Between 18 and 65 years | 0 | 0 | 0
  Participants under 18 years: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 142 | 140 | 282
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 142 | 136 | 278
  Coloured | 0 | 1 | 1
  Other | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  South Africa | 142 | 140 | 282

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Expressed Satisfaction With the Intervention
Description: Client Satisfaction Questionnaire - Using the client satisfaction questionnaire, investigators will measure satisfaction using likert scale responses that range from 1 to 5 with 5 aligning with high satisfaction with the intervention. Investigators are aiming for 80% of more of participants with rankings of satisfied or higher. The questionnaire is based off of the following measure: Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: Development of a general scale. Evaluation and Program Planning. 1979;2:197-207.
  Only participants in the intervention arm answer questions on satisfaction with the intervention.
Time Frame: 6 months
Population: Participants assigned to the intervention arm, and who were exposed to the experimental intervention, answered questions on satisfaction with the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 140
Participants | 113

2. Primary Outcome: Number of Participants Who Were Retained At the 6-month Time Point
Description: There is no scale for feasibility. Investigators will look at retention rates. Feasibility will be aligned with 75% or higher retention rates at the 6 month timepoint.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 142 | 140
Participants | 140 | 139

3. Secondary Outcome: Prevention or Reduction of Sexual Behavior Related to HIV Acquisition Risk as Measured Through the Percent of Participants Engaged in Lifetime Condom Use.
Description: This is an underpowered outcome because the primary goal of this study is not to evaluate efficacy. There is no scale for these behaviors. For this secondary outcome, investigators will examine the percent of participants who engaged in lifetime condom use. This will be reported for each arm, comparing percentages engaged in lifetime condom use at the 6-month time point for each arm separately.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 142 | 140
Participants
  Number of participants engaged in lifetime condom use at 1 month | 95 | 92
  Number of participants engaged in lifetime condom use at 6 months | 98 | 99

4. Secondary Outcome: Prevention or Reduction of Attempted or Completed Acts of Intimate Partner Violence Using Mary Koss's Short Form Sexual Violence Perpetration Scale At the 1-month Time Point
Description: This is an underpowered outcome because the primary goal of this study is not to evaluate efficacy. For this secondary outcome, investigators will examine if there is a decrease in incidents of attempted and completed acts of sexual violence. The percentage of participants engaged in any completed act of sexual perpetration - defined as 1 or more acts of forced touching, oral sex, anal sex, and/or vaginal sex - will be compared for the intervention arm, looking at baseline versus 1 month. Similarly, the percentage of participants engaged in any completed act of sexual perpetration - defined as 1 or more acts of forced touching, oral sex, anal sex, and/or vaginal sex - will be compared for the control arm, looking at baseline versus 1 month.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 142 | 140
Participants | 78 | 81

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from the date of enrollment until 6 month followup (the last followup timepoint).
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/142 | 1/140
Serious Adverse Events (participants affected / at risk) | 0/142 | 1/140
Other Adverse Events (participants affected / at risk) | 0/142 | 0/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=142) | Control (N=140)
Death of study participant (General disorders) | 0 (0) | 1 (1) — A study participant died prior to completion of the 6 month follow-up survey. The participant died due to a headache not connected to study procedures. The IRB reviewed this incident and determined that this death was not study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT05869864/Prot_SAP_001.pdf